CLINICAL TRIAL: NCT04282668
Title: A Phase 1 Study of Safety, Pharmacokinetics, and Preliminary Activity of TAS1440, as a Single Agent and in Combination With All-Trans Retinoic Acid (ATRA) in Subjects With Relapsed or Refractory (r/r) Acute Myeloid Leukemia (AML)
Brief Title: A Study of TAS1440 With ATRA in Subjects With r/r AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to the changing treatment landscape, difficulty in enrolling eligible participants, and little likelihood of providing meaningful clinical benefit for the participants.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAS1440-01
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAS1440 (Experimental): TAS1440 as a single agent administered once daily (QD) on specific days during each 28-day cycle in Part 1.
  Interventions: Drug: TAS1440
- TAS1440 + ATRA (Experimental): TAS1440 administered QD on specific days during each 28-day cycle in combination with ATRA twice daily (BID) in Part 2.
  Interventions: Drug: TAS1440 + ATRA

INTERVENTIONS:
Drug: TAS1440 — Form: Capsule or Tablet Route of Administration: Oral
  Arms: TAS1440
Drug: TAS1440 + ATRA — Form: Capsule or Tablet Route of Administration: Oral
  Other Names: Tretinoin; Vesanoid
  Arms: TAS1440 + ATRA

SUMMARY:
This is a multicenter, 2-part, Phase 1 study to assess the safety, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of TAS1440 administered as a single agent and in combination with all-trans retinoic acid (ATRA) in participants with acute myeloid leukemia (AML) who have relapsed or are refractory (r/r) to prior treatment. The study duration is expected to be approximately 30 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have a projected life expectancy of at least 12 weeks and be in stable condition to complete 1 full cycle (4 weeks) of treatment.
2. Have histological confirmation of AML by World Health Organization (WHO) 2016 criteria and who have failed all other available conventional therapies.
3. Have a peripheral blood or bone marrow blast count >5% at the time of enrollment.
4. Have disease that:

   1. is refractory to standard induction chemotherapy, including but not limited to anthracycline and cytarabine combination therapy, or
   2. has relapsed after anthracycline and cytarabine therapy or stem cell transplant (SCT), or
   3. is refractory to or has relapsed after a front-line regimen containing a hypomethylating agent, alone or in combination.
5. Have an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 1.
6. Have adequate renal function as demonstrated by a serum creatinine ≤1.5 × upper limit of normal (ULN) or calculated creatinine clearance (by the standard Cockcroft-Gault formula) of ≥60 mL/min.
7. Have adequate liver function as demonstrated by the following:

   1. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × upper limit of normal (ULN)
   2. AST and ALT <5 × ULN (if considered due to leukemic organ involvement).
8. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Known clinically active central nervous system leukemia.
2. BCR-ABL-positive leukemia.
3. Diagnosis of acute promyelocytic leukemia (M3 AML or APML or APL).
4. Second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy.
5. Grade 3 or higher graft versus host disease (GVHD), or GVHD requiring treatment with either:

   1. a calcineurin inhibitor, or
   2. prednisone more than 5 mg/day (Note: Prednisone at any dose for other indications is allowed).
6. Total serum bilirubin ≥1.5 × ULN (except for subjects with Gilbert's Syndrome for whom direct bilirubin is >2.5 × ULN), or liver cirrhosis, or chronic liver disease Child-Pugh Class B or C.
7. Known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status or low viral hepatitis titer being treated with antivirals is allowed. For subjects considered at risk of viral exposure, serologies should be used to establish negativity.
8. Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the subject to high risk of non-compliance with the protocol.
9. Myocardial impairment of any cause (eg, cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, or congestive heart failure) resulting in heart failure by New York Heart Association (NYHA) Criteria (Class III or IV staging).
10. Screening 12-lead echocardiogram with measurable QTc interval (according to either Fridericia's or Bazett's correction) of >480 milliseconds.
11. Active, uncontrolled infection. Participants with an infection receiving treatment (antibiotic, antifungal, or antiviral treatment) must be afebrile and hemodynamically stable for ≥72 hours before enrollment.
12. Non-AML-associated pulmonary disease requiring >2 liters per minute (LPM) oxygen.
13. Proliferative AML with total white blood cells > 20,000/uL
14. Any other condition that puts the participant at an imminent risk of death.
15. Treated with any investigational therapy within 2 weeks of the first dose of study treatment.
16. Inability to swallow oral medication.
17. Known hypersensitivity to ATRA, any of its components, or other retinoids.
18. Known sensitivity to parabens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Safety: Number of participants with treatment-emergent adverse events (TEAEs) | Approximately 30 months

SECONDARY OUTCOMES:
Response rate: Number of participants with complete remission (CR), complete remission with incomplete blood count recovery (CRi), partial remission (PR) and complete remission with partial hematological recovery (CRh) | Approximately 30 months
Overall survival: Time from the date of the first dose until death due to any cause | Approximately 30 months
Pharmacokinetic parameter: Area under the curve (AUC) | Up to Day 8 of Cycle 1 and Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Maximum plasma concentration (Cmax) | Up to Day 8 of Cycle 1 and Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Minimum plasma concentration (Cmin) | Up to Day 8 of Cycle 1 and Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Time to reach maximum plasma concentration (Tmax) | Up to Day 8 of Cycle 1 and Cycle 2 (28 days per cycle)
Pharmacokinetic parameter: Half-life (t1/2) | Up to Day 8 of Cycle 1 and Cycle 2 (28 days per cycle)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Arizona Cancer Center Site#127, Tucson, Arizona
  - Norton Cancer Institute Site# 108, Louisville, Kentucky
  - University of Michigan Medical School Site#107, Ann Arbor, Michigan
  - Oregon Health and Science University Site#111, Portland, Oregon
  - Fox Chase Cancer Center Site#112, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute Site#110, Dallas, Texas
  - MD Anderson Cancer Center Site#101, Houston, Texas
  - Fred Hutchinson Cancer Research Center Site#105, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No